CLINICAL TRIAL: NCT00526747
Title: Novel Biomarkers of Erythropoietin Resistant Anemia Among Patients With Chronic Kidney Disease
Brief Title: Erythropoietin Resistance in Anemia of Chronic Kidney Disease
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00008469
Record Dates: First submitted 2007-09-06; First posted 2007-09-10 (Estimated); Last update posted 2013-04-11 (Estimated); Status verified 2008-11

CONDITIONS: Anemia; Kidney Failure; Erythropoietin
MeSH Terms: conditions — Anemia; Renal Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Epo-resistant: Patients with CKD (estimated GFR < 60cc/min) not on hemodialysis who are receiving greater than or equal to 100IU/kg/week of epoetin alpha and/or 1mcg/kg/week darbepoetin to obtain target hemoglobin or hematocrit.
- Epo-responsive: Patients with CKD (estimated GFR < 60cc/min) not on hemodialysis who are requiring <100IU/kg/week of epoetin alpha and/or 1mcg/kg/week of darbepoetin to obtain target hemoglobin/hematocrit.

SUMMARY:
Our goal of this pilot project is to identify inflammatory biomarkers that correlate with epo-resistance among CKD patients.

ELIGIBILITY:
Inclusion Criteria:

* prevalent patients greater than or equal to 18 years old with CKD defined as a glomerular filtration rate < 60 cc/min

Exclusion Criteria:

* active GI bleeding or history of GI bleed in the prior 3 months
* uncontrolled hyperparathyroidism (PTH>500)
* untreated iron deficiency (transferrin saturation < 20% and ferritin < 100
* overt infection
* active hemolysis
* hemoglobinopathies
* known adverse response to erythropoietin
* prior kidney transplant
* aluminum toxicity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: CKD anemia clinic patients
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2007-08; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jula Inrig, MD, MHS, Principal Investigator — Duke University; Lynda Szczech, MD, Principal Investigator — Duke University; Suzanne K Bryskin, MD, Principal Investigator — Duke University
Locations (2):
- United States (2):
  - Durham Nephrology Anemia Clinic, Durham, North Carolina
  - Duke University Medical Center Anemia Clinic, Durham, North Carolina

REFERENCES:
- [Background] Rossert J, Gassmann-Mayer C, Frei D, McClellan W. Prevalence and predictors of epoetin hyporesponsiveness in chronic kidney disease patients. Nephrol Dial Transplant. 2007 Mar;22(3):794-800. doi: 10.1093/ndt/gfl716. Epub 2007 Jan 8. PMID 17210593
- [Background] McClellan WM, Flanders WD, Langston RD, Jurkovitz C, Presley R. Anemia and renal insufficiency are independent risk factors for death among patients with congestive heart failure admitted to community hospitals: a population-based study. J Am Soc Nephrol. 2002 Jul;13(7):1928-36. doi: 10.1097/01.asn.0000018409.45834.fa. PMID 12089390
- [Background] U.S. Renal Data System, USRDS 2005 Annual Data Report: Atlas of End-Stage Renal Disease in the United States, National Institutes of Health, National Institutes of Diabetes and Digestive and Kidney Disease, Bethesda, MD, 2005.
- [Background] McMahon LP, Mason K, Skinner SL, Burge CM, Grigg LE, Becker GJ. Effects of haemoglobin normalization on quality of life and cardiovascular parameters in end-stage renal failure. Nephrol Dial Transplant. 2000 Sep;15(9):1425-30. doi: 10.1093/ndt/15.9.1425. PMID 10978402
- [Background] Evans RW, Rader B, Manninen DL. The quality of life of hemodialysis recipients treated with recombinant human erythropoietin. Cooperative Multicenter EPO Clinical Trial Group. JAMA. 1990 Feb 9;263(6):825-30. PMID 2404150
- [Background] Wolcott DL, Marsh JT, La Rue A, Carr C, Nissenson AR. Recombinant human erythropoietin treatment may improve quality of life and cognitive function in chronic hemodialysis patients. Am J Kidney Dis. 1989 Dec;14(6):478-85. doi: 10.1016/s0272-6386(89)80148-9. PMID 2596475
- [Background] Strippoli GF, Craig JC, Manno C, Schena FP. Hemoglobin targets for the anemia of chronic kidney disease: a meta-analysis of randomized, controlled trials. J Am Soc Nephrol. 2004 Dec;15(12):3154-65. doi: 10.1097/01.ASN.0000145436.09176.A7. PMID 15579519
- [Background] Obrador GT, Roberts T, St Peter WL, Frazier E, Pereira BJ, Collins AJ. Trends in anemia at initiation of dialysis in the United States. Kidney Int. 2001 Nov;60(5):1875-84. doi: 10.1046/j.1523-1755.2001.00002.x. PMID 11703606
- [Background] Zhang Y, Thamer M, Stefanik K, Kaufman J, Cotter DJ. Epoetin requirements predict mortality in hemodialysis patients. Am J Kidney Dis. 2004 Nov;44(5):866-76. PMID 15492953
- [Background] Humphries JE. Anemia of renal failure. Use of erythropoietin. Med Clin North Am. 1992 May;76(3):711-25. doi: 10.1016/s0025-7125(16)30349-2. PMID 1578966
- [Background] Stenvinkel P. Anaemia and inflammation: what are the implications for the nephrologist? Nephrol Dial Transplant. 2003 Nov;18 Suppl 8:viii17-22. doi: 10.1093/ndt/gfg1086. PMID 14607995
- [Background] Kimmel PL, Phillips TM, Simmens SJ, Peterson RA, Weihs KL, Alleyne S, Cruz I, Yanovski JA, Veis JH. Immunologic function and survival in hemodialysis patients. Kidney Int. 1998 Jul;54(1):236-44. doi: 10.1046/j.1523-1755.1998.00981.x. PMID 9648084
- [Background] Macdougall IC, Cooper AC. Erythropoietin resistance: the role of inflammation and pro-inflammatory cytokines. Nephrol Dial Transplant. 2002;17 Suppl 11:39-43. doi: 10.1093/ndt/17.suppl_11.39. PMID 12386257
- [Background] Nemeth E, Rivera S, Gabayan V, Keller C, Taudorf S, Pedersen BK, Ganz T. IL-6 mediates hypoferremia of inflammation by inducing the synthesis of the iron regulatory hormone hepcidin. J Clin Invest. 2004 May;113(9):1271-6. doi: 10.1172/JCI20945. PMID 15124018
- [Background] Bologa RM, Levine DM, Parker TS, Cheigh JS, Serur D, Stenzel KH, Rubin AL. Interleukin-6 predicts hypoalbuminemia, hypocholesterolemia, and mortality in hemodialysis patients. Am J Kidney Dis. 1998 Jul;32(1):107-14. doi: 10.1053/ajkd.1998.v32.pm9669431.
- [Background] Sitter T, Bergner A, Schiffl H. Dialysate related cytokine induction and response to recombinant human erythropoietin in haemodialysis patients. Nephrol Dial Transplant. 2000 Aug;15(8):1207-11. doi: 10.1093/ndt/15.8.1207. PMID 10910446
- [Background] Touam M, Guery B, Goupy C, Menoyo V, Drueke T. Hypothyroidism and resistance to human recombinant erythropoietin. Nephrol Dial Transplant. 2004 Apr;19(4):1020-1. doi: 10.1093/ndt/gfg556. No abstract available. PMID 15031379
- [Background] Danielson B. R-HuEPO hyporesponsiveness--who and why? Nephrol Dial Transplant. 1995;10 Suppl 2:69-73. doi: 10.1093/ndt/10.supp2.69. PMID 7644109
- [Background] Goicoechea M, Martin J, de Sequera P, Quiroga JA, Ortiz A, Carreno V, Caramelo C. Role of cytokines in the response to erythropoietin in hemodialysis patients. Kidney Int. 1998 Oct;54(4):1337-43. doi: 10.1046/j.1523-1755.1998.00084.x. PMID 9767553
- [Background] Nemeth E, Tuttle MS, Powelson J, Vaughn MB, Donovan A, Ward DM, Ganz T, Kaplan J. Hepcidin regulates cellular iron efflux by binding to ferroportin and inducing its internalization. Science. 2004 Dec 17;306(5704):2090-3. doi: 10.1126/science.1104742. Epub 2004 Oct 28. PMID 15514116
- [Derived] Inrig JK, Bryskin SK, Patel UD, Arcasoy M, Szczech LA. Association between high-dose erythropoiesis-stimulating agents, inflammatory biomarkers, and soluble erythropoietin receptors. BMC Nephrol. 2011 Dec 12;12:67. doi: 10.1186/1471-2369-12-67. PMID 22152013